CLINICAL TRIAL: NCT03324490
Title: Comparative Study of Mid-thoracic Spinal Versus Epidural Anesthesia for Open Nephrectomy in Patients With Obstructive/Restrictive Lung Disease: A Randomized Controlled Study
Brief Title: Thoracic Spinal Versus Epidural Anesthesia for Nephrectomy in Obstructive/Restrictive Lung Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TSEANORLDP60
Record Dates: First submitted 2017-10-18; First posted 2017-10-27 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Nephrectomy; Lung Diseases; Anesthesia
Keywords: Mid-thoracic spinal anesthesia; Mid-thoracic epidural anesthesia; Nephrectomy; Lung disease
MeSH Terms: conditions — Lung Diseases | interventions — Bupivacaine; Fentanyl; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Using computer & sealed envelope randomization, patients are assigned to receive either thoracic spinal anesthesia [TSA group: n=30] or thoracic epidural anesthesia [TEA group: n=30].
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TSA group (Active Comparator): Thoracic Spinal Anesthesia; Bupivacaine 0.5% (hyperbaric) 7.5mg, Fentanyl 25 µg & Dexmedetomidine 5 µg by intrathecal injection
  Interventions: Procedure: Thoracic Spinal Anesthesia; Drug: Bupivacaine 0.5% (hyperbaric); Drug: Fentanyl; Drug: Dexmedetomidine
- TEA group (Active Comparator): Thoracic Epidural Anesthesia; Bupivacaine 0.5% (isobaric) 25-50 mg & Fentanyl 10-20 µg by epidural injection
  Interventions: Procedure: Thoracic Epidural Anesthesia; Drug: Bupivacaine 0.5% (isobaric); Drug: Fentanyl

INTERVENTIONS:
Procedure: Thoracic Spinal Anesthesia — Spinal anesthesia will be performed for patients of the TSA group at the T7-T8 intervertebral space, using a 27 G pencil point needle with an introducer (Braun Melsungen, Melsungen, Germany).
  When correct placement is confirmed by the free flow of clear CSF, 1.5 ml of hyperbaric Bupivacaine 0.5% (7.5 mg) in addition to 0.5 ml Fentanyl (25 μg) & 5 μg dexmedetomidine will be injected.
  Arms: TSA group
Procedure: Thoracic Epidural Anesthesia — Epidural anesthesia will be performed for patients of the TEA group at the T7-T8 intervertebral space, using the "Prefix Custom Epidural Anesthesia Tray" with an 18 G Tuohy epidural needle & a 20 G epidural catheter.
  Patients will initially receive 5-10 ml of a mixed preparation of 0.5% isobaric Bupivacaine with 2 μg Fentanyl per ml volume as a bolus dose via the epidural catheter, this will be followed by a continuous infusion of 5-10 ml/hr started 1 hour after the bolus dose & continued throughout the procedure.
  Arms: TEA group
Drug: Bupivacaine 0.5% (hyperbaric) — Neuro-axially injected
  Other Names: Heavy Marcaine
  Arms: TSA group
Drug: Bupivacaine 0.5% (isobaric) — Neuro-axially injected
  Other Names: Marcaine
  Arms: TEA group
Drug: Fentanyl — Neuro-axially injected
Drug: Dexmedetomidine — Neuro-axially injected
  Arms: TSA group

SUMMARY:
Patients with respiratory disease have an increased risk of developing complications perioperatively. The use of regional anesthesia decreases this risk with better postoperative outcome. The aim of this study is to compare the safety and efficacy of thoracic spinal versus thoracic epidural anesthesia for open nephrectomy in patients with obstructive/restrictive lung disease.

ELIGIBILITY:
Inclusion Criteria:

* ASA class II or III
* Mild to moderate obstructive or restrictive lung disease
* Open nephrectomy candidate patients

Exclusion Criteria:

* Any condition contra-indicating regional anesthesia
* Allergic to any of the drugs used during the procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction Score | 24 hours
  Patient Satisfaction Score defines the degree of patient satisfaction with the anesthetic experience and is assessed after recovery. It is graded as excellent "E" (best score), fair "F" & poor "P" (worst score).

SECONDARY OUTCOMES:
VAS | 12 hours
  Visual Analogue Score for pain graded from 0-10 [0: no pain, 10: worst pain].
Mean ABP | 12 hours
  Change in Mean Arterial Blood Pressure measured in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Nazmy E Seif, MD, Study Chair — Kasr Al-Ainy Hospital, Cairo University; Ahmed M El-Badawy, MD, Study Director — Kasr Al-Ainy Hospital, Cairo University
Locations (1):
- Kasr Al-Ainy Hospital, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided